CLINICAL TRIAL: NCT07027124
Title: Neoadjuvant ADT and Darolutamide With Pembrolizumab, Followed by Adjuvant Pembrolizumab in NCCN High-risk and Molecularly Stratified Prostate Cancer Patients
Brief Title: Neoadjuvant ADT + Darolutamide With Pembrolizumab, Followed by Adjuvant Pembrolizumab in Molecularly Stratified High-Risk Prostate Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Bayer (Industry)
Responsible Party: Principal Investigator, Ashutosh Kumar Tewari, Urology Chair, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-23-01400
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; High-risk Prostate Cancer
Keywords: Prostate Cancer; Immunotherapy; Pembrolizumab; Darolutamide; ADT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; pembrolizumab; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with Prostate Cancer (Experimental): Neoadjuvant ADT plus AR- antagonist, Darolutamide plus Pembrolizumab (5 cycles) prior to radical prostatectomy (RP) in a stratified high-risk localized prostate cancer cohort, followed by adjuvant treatment with Pembrolizumab (12 cycles) post-RP.
  Interventions: Drug: Darolutamide; Drug: Pembrolizumab; Drug: Lupron

INTERVENTIONS:
Drug: Darolutamide — Darolutamide 600 mg (2 tablets of 300 mg) twice daily with food, equivalent to a total daily dose of 1200 mg for 16 weeks prior to RP.
  Other Names: Nubeqa
Drug: Pembrolizumab — Administered at the dose of 200 mg intravenously, every 3 weeks, for a total of 5 cycles prior to RP (Neoadjuvant phase, study weeks 1, 4, 7, 10, 13 & 16), and every 3 weeks, for a total of 12 cycles post-RP (Adjuvant phase, study weeks, 19, 22, 25, 28, 31, 34, 37, 40 43, 46, 49, & 52). Total Pembrolizumab cycles=17
  Other Names: Keytruda
Drug: Lupron — Androgen deprivation, GnRH agonist Leuprolide will be administered at a dose of 22.5 mg SQ (Eligard)/IM Lupron every 12 weeks prior to RP (Study weeks, 1 and 13).
  Other Names: Leuprolide

SUMMARY:
This is a single-arm, phase II study of neoadjuvant combination therapy of Androgen Deprivation Therapy (ADT), [Gonadotropin-Releasing Hormone (GnRH) agonist Leuprolide], androgen receptor (AR)-antagonist Darolutamide and Pembrolizumab in a stratified high-risk localized prostate cancer cohort, followed by adjuvant treatment with Pembrolizumab (12 cycles) post-radical prostatectomy (RP).

Patients with National Comprehensive Cancer Network (NCCN) high-risk non-metastatic prostate cancer (localized or locally advanced) (defined as Gleason ≥8, disease stage >=cT3a, or PSA l >20 ng/mL) will be risk-stratified at a biopsy using Decipher, a commercial standard-of-care diagnostic assay. Patients satisfying all three criteria of high-risk genomic characteristics listed below as per the Decipher grid results will be enrolled in the study:

1. Decipher Genomic classifier, GC>0.6
2. AR activity score/AR-output gene signature (ARoS)>11.0
3. High Luminal B score/ PAM50 subtype signature

DETAILED DESCRIPTION:
The objectives of this study are to evaluate if the neoadjuvant ADT, Darolutamide and Pembrolizumab treatment in high-risk prostate cancer patients stratified based on their genomic characteristics will lead to minimum residual disease (MRD).

A total of 40 men ≥ 18 years of age with non-metastatic adenocarcinoma of the prostate, having NCCN high risk localized disease, risk stratified at biopsy based on Decipher score, AR activity score and Luminal B score will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male Age ≥ 18 years at the time of consent
* Patients must have histopathologically confirmed adenocarcinoma of the prostate
* Patients must have NCCN high-risk localized or locally advanced prostate cancer and absence of distant metastasis or nodal involvement defined as those having one of the following.

  * Gleason score ≥ 8
  * PSA > 20 ng/ml
  * Clinical stage >cT2C (T3a and above)
* Patients must be risk-stratified at biopsy and their cancer should have all three molecular features given below at baseline.

  * Decipher Genomic Classifier >0.6 (interpreted from decipher report)
  * High AR activity/AR activity score >11 (interpreted from decipher report)
  * Luminal B subtype (interpreted from decipher report)
* The patient must have a performance status of 0-1 as determined by criteria set forward by the eastern cooperative oncology group.
* Patients with prior neoadjuvant hormonal therapy are allowed if they meet the following criteria.

  * have completed all treatments ≥ 12, months ago.
  * Recovered from all AEs due to previous therapies.
* If patient has had a major surgery, he should have recovered from all complications and toxicities prior to enrolling in the study.
* Adequate organ and marrow function as defined below:

  * Hematological
  * Absolute neutrophil count (ANC) ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcl
  * Hemoglobin (Hb) ≥ 9 g/dL Hepatic
  * total bilirubin ≤ 1.5 mg/dl (except in patients with gilbert syndrome who can have total bilirubin <3.0 mg/dl)
  * Aspartate aminotransferase (AST) ≤ 2.5 x ULN
  * Alanine aminotransferase (ALT) ≤ 2.5 x ULN Renal
  * Creatinine OR Creatinine ≤ 1.5 ULN OR
  * Calculated creatinine clearance Creatinine clearance ≥ 30 ml/min
  * Men must agree to use a condom and not father a child or donate sperm for the duration of the study and for 90 days after completion of therapy. Subject must agree to partner use of an additional contraceptive method when having intercourse with women of childbearing potential (WOCBP).
  * Ability to understand and the willingness to sign a written informed consent.
  * Participants who are HBs Ag positive are eligible if they have received HBV anti-viral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.

Note: Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.

* Hepatitis B screening tests are not required unless:

  * Known history of HBV infection
  * As mandated by local health authority
* Participants with a history of HCV infection are eligible if HCV viral load is undetectable at screening.

Note: Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.

* Hepatitis C screening tests are not required unless:

  * Known history of HCV infection
  * As mandated by local health authority
* Participants with a known history of Human immunodeficiency virus (HIV) infection are eligible as long as they have an undetectable viral. HIV positive participants must be taking stable ART for ≥ 12 weeks and have an undetectable HIV viral load within 28 days before enrollment. Minor fluctuations up to 200 copies/mL are acceptable.

Exclusion Criteria:

* Patients with metastatic disease
* Patients with Gleason score <8
* Patients with Biopsy Decipher score ≤0.6.
* Patients have had prior hormonal therapy (please see inclusion criteria for exceptions).
* Patients have had prior radiation therapy or chemotherapy for prostate cancer.
* Patients with active cardiac disease defined as having any of the following within 6 months prior to the start of treatment:

  * myocardial infarction,
  * severe/unstable angina pectoris,
  * congestive heart failure,
  * hospitalization for any cardiac event
* Patients has active GI disorder that will interfere with absorption of study drug Darolutamide Subject has prior treatment with androgen receptor inhibitors, such as apalutamide, Darolutamide, enzalutamide, abiraterone acetate or other investigational CYP17 inhibitor.
* Inability to swallow oral medications.
* Patients has active infection requiring systemic therapy within 7 days of Week 1.
* Patients has received prior therapy with anti-PD1, anti-PDL1, anti-PDL2 or with other checkpoint inhibitors or T-cell costimulatory/inhibitory agents (e.g., CD137, OX-40, CTLA4).
* Patients with an active viral Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive or detectable [qualitative] Hepatitis b virus [HBV] DNA or defined as Hepatitis V virus [HCV] ribonucleic acid [RNA] [qualitative] is detected), known Human Immunodeficiency virus (HIV) infection with detectable viral load, or chronic liver disease with a need of treatment.
* Patients has a known active or known history of TB (Bacillus tuberculosis) or active history of non-infectious pneumonitis.
* Patients who are immunodeficient or are receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days of study intervention. Topical or inhaled steroids are permitted in absence of immunodeficiency or autoimmune disease.
* Patients have active auto-immune disease that has required systemic therapy (use of disease modifying agents, corticosteroids, or immunosuppressive drugs) in the past 2 years. However, subjects receiving replacement therapy (e.g., insulin, thyroxine, or physiological corticosteroid replacement therapy for adrenal and pituitary insufficiency) are eligible.
* Has history or current evidence of any condition, therapy that might confound results of the study. - Has known psychiatric, epileptic or substance abuse history or disorder that would interfere with participant's ability to cooperate with the requirements of the study.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Known history of allergic reactions attributed to compounds of similar chemical or biologic composition to Agent(s) or other agents used in study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer Patients
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2031-05-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve Minimal residual disease (MRD) | at time of surgery (At Week 17)
  MRD is defined as residual cancer burden (RCB) ≤0.25cm³ at final pathology, where RCB is calculated by multiplying the residual tumor volume with the tumor cellularity. The proportion of patients who achieve MRD will be collected at the time of surgery.

SECONDARY OUTCOMES:
Complete pathological response (pCR) | After Week 17
  Complete pathological response (pCR) is defined as the absence of viable tumor in post treatment prostatectomy specimens). pCR is typically determined by examining the radical prostatectomy specimen after surgery.
Proportion of patients who had had their tumor downstaged | at time of surgery (At Week 17)
  Proportion of patients who had had their tumor downstaged due to neoadjuvant Pembrolizumab, Darolutamide and ADT at the time of surgery. Downstaging will be determined using MRI and pathology separately.
Adverse events assessed by NCI CTCAE (v.5.0). | Week 1 to Week 16, Week 19 to Week 52
  Adverse events assessed by NCI CTCAE (v.5.0). Incidence of AEs will be reported for the first cycle of neoadjuvant therapy, for the entire neoadjuvant treatment phase, and for the adjuvant treatment phase.
Biochemical progression free survival bPES | Week 22 and until 5 years after Week 17
  bPFS is defined as the time from baseline to first evidence of biochemical progression based on PSA level or death, whichever occurs first.
Metastasis free survival (MFS) | Week 17 and until 5 years after Week 17
  Metastasis free survival (MFS) defined as time from enrollment to detection of metastasis or death, whichever occurs first.
Tumor Volumes | Week 0 to Week 17
  Median tumor volumes assessed by MRI at baseline and before surgery (and the corresponding change in median tumor volume from baseline to before surgery).
Immunological responses in blood | Week 0 to Week 52
  A broad immunophenotyping panel will be used to define various immune subsets and their functional states, in pre-treatment and longitudinally collected whole blood samples. Longitudinally collected serum/plasma samples will be analyzed using Olink multiplex assay platform.
Whole exome-sequencing (WES) | Week 0 to Week 17
  Transcriptomic and genomic changes in tissues - Whole exome-sequencing (WES) will be performed for characterization of the mutational landscape including neoantigens and differentially expressed genes and gene signatures.
RNA sequencing (RNA-seq) | Week 0 to Week 17
  Transcriptomic and genomic changes in tissues - RNA sequencing (RNA-seq) will be performed for characterization of the mutational landscape including neoantigens and differentially expressed genes and gene signatures.

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh K Tewari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Dimple Chakravarty, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis.
  Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in ISMMS data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be determined).